CLINICAL TRIAL: NCT00003207
Title: Phase I Study on Doxil and SDZ PSC 833 in the Treatment of AIDS-Associated Kaposi's Sarcoma and Other Advanced Malignancies
Brief Title: Liposomal Doxorubicin and PSC 833 in Treating Patients With AIDS-Related Kaposi's Sarcoma or Other Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000066062; WU-106; NCI-T97-0073
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Sarcoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — liposomal doxorubicin; valspodar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 1 (Doxil & PSC 833) (Experimental): Patients will receive Doxil at the standard dose of 20 mg/m2 IV for the 1st cycle. On the 2nd cycle of Doxil, the first patient will receive Doxil at 40% of standard dose or 8 mg/m2 (dose level 1) IV over one hr. 15 mn after the 2nd and subsequent cycles of Doxil, PSC 833 will be given at 2 mg/kg for 2 hrs. Simultaneously, a 72 hour CIVI of PSC 833 will be started with the loading dose. If no DLT occurs, then a double dose escalation of Doxil (dose levels 3, 5, 7 ) will be given to the same patient in the subsequent cycles until DLT occurs. On the 2nd cycle, Doxil will be given at the next dose level above the starting dose tolerated by the first patient. If no DLT occurs, a double dose escalation will also be done for the subsequent cycles (dose levels 5, 7, 9). The single-patient-cohort will terminate when a patient experiences DLT or when two episodes of grade 2 toxicity occur. At that point patients will be enrolled into cohorts of 3 patients to determine the MTD.
  Interventions: Drug: pegylated liposomal doxorubicin hydrochloride; Drug: PSC 833

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride
  Other Names: DOXIL
Drug: PSC 833
  Other Names: valspodar

SUMMARY:
The rationale for conducting this study lies in the premise that if indeed the reason for a limited response of Kaposi's sarcoma lesions and other advanced malignancies to chemotherapy is attributable to a high expression of P-glycoprotein, then, by inhibiting this pump, tumor kill would be enhanced and response rates as well as duration of responses would also increase. Doxil is chosen since recent studies have shown that it is superior to combination chemotherapy with ABV or BV. Doxil is also known to be active in other malignancies such as breast and ovarian cancer (34,35). PSC 833 is chosen since it has been found to reverse P-gp in vitro and in vivo, is non-immunosuppressive, and has been shown in recent Phase 1 studies to be well tolerated.

There are yet no human studies reported on Doxil pharmacokinetics when combined with MDR modulators. Preclinical data shows that pharmacokinetics of Doxil, unlike free doxorubicin, is minimally affected by the addition of PSC 833 (36). Enhanced tumor toxicity was observed when PSC 833 was combined with Doxil. Since doxorubicin, the active agent in Doxil, is metabolized by the same cytochrome P450, interactions between these 2 agents may have very significant clinical implications. The purpose of this study is to assess the toxicity and determine the maximum tolerated dose of Doxil when combined with PSC 833 in the treatment of AIDS-KS and other advanced malignancies.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically documented malignancy refractory to standard treatment or for which no standard treatment exists, or biopsy proven Kaposi's sarcoma with mucocutaneous lesions numbering 10 or more or a documented visceral KS lesion with at least 2 assessable cutaneous lesions.
* A life expectancy of >4 months.
* Patients with prior chemotherapy and Doxil exposure are eligible
* Age >=18
* Karnofsky score of >=70%
* Hemoglobin >=8 g/dl, neutrophil count >=1000 cells/ul and platelet count of >=75,000 cells/ul.
* Creatinine clearance of .=50 ml/min or creatinine of <=2.0mg/dl, SGOT <=2X the institutional normal and bilirubin <1.5X institutional normal
* Written informed consent has been obtained from the patient.

EXCLUSION CRITERIA

* Pregnant or breast feeding patients as radioactive tracer material and chemotherapy will be used in this protocol.
* Active opportunistic infections requiring antibiotic treatment.
* Treatment with radiation or electron beam therapy, interferon or cytotoxic therapy within the preceding 4 weeks.
* Clinically significant history of congestive heart failure.
* Patients who have moderate to severe sensory and motor peripheral neuropathy.
* Any patient currently receiving treatment with any of the following agents which cannot be discontinued at a specified time relative to PSC 833 administration. All of these drugs are well substantiated to interact with cyclosporin A:

  * Agents increasing serum concentrations of CsA

The following drugs must not be administered for 48 hours before PSC 833 is started, during the course of its administration, or up to 48 hours after the last dose of PSC 833 in a cycle:

Calcium channel blockers: diltiazem, nicardipine, verapamil Antifungals: fluconazole (dose <200 mg/day allowed), itraconazole, ketoconazole Antibiotics: clarithromycin, erythromycin Others: metoclopramide,bromocriptine, danazol

* Agents decreasing serum concentrations of CsA

The following drugs must not be administered in the 14 days before PSC 833 is started or during the course of its administration. They may be restarted immediately after the last dose of PSC 833:

Antibiotics: nafcillin, rifampin Anticonvulsants: carbamazepine, phenobarbital, phenytoin Others: octreotide, ticlopidine

* Hypersensitivity to Doxil or cyclosporin A
* Any patient, who, in the judgment of the investigator, may not be able to complete this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1998-03; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Safety profile and tolerability of Doxil in combination with PSC 833
  Each cycle is 2 weeks long and can continue until disease progression, toxicity, or patient decision
Maximum tolerated dose of Doxil in combination with PSC 833
Dose limiting toxicity of Doxil in combination with PSC 833

SECONDARY OUTCOMES:
Effects of PSC 833 on Doxil pharmacokinetics
Confirm the MDR expression with immunohistochemistry and functionally, with 99MTc-sestamibi

CONTACTS AND LOCATIONS:
Overall Officials: Paula M. Fracasso, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States